CLINICAL TRIAL: NCT05274152
Title: Immersive Virtual Reality: Lower Limb and Knee Rehabilitation in Young People
Brief Title: Using Immersive Virtual Reality for Children's Lower Limb Rehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheffield Hallam University (Other)
Collaborators: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: AA14737018
Record Dates: First submitted 2022-03-01; First posted 2022-03-10 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Virtual Reality; Physical Rehabilitation; Lower Limb Injury; Paediatric
MeSH Terms: conditions — Leg Injuries

STUDY DESIGN:
Intervention Model Description: The study will take the form of feasibility and proof of concept trial using IVR as a physiotherapy rehabilitation tool following lower limb or knee surgery for children (aged 11 - 16). It will examine the feasibility, acceptability, usability, and efficacy of the IVR system from the perspectives of the children, parents and staff. The mixed-method approach (collecting quantitative and qualitative data)
  Participants:
  Child participants (n=15) will be patients of Sheffield Teaching Hospitals NHS Trust.
  Inclusion criteria, aged 11-16.
  This study also included parents who have child participating in the study and being able to speak and understand English.; and physiotherapists involved in the physical therapeutic. There are no exclusion criteria for parents or staff, so long as they meet the inclusion criteria.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients IVR for Lower Limb and Knee Rehabilitation after surgery in children (Experimental): Patients will use the IVR during each physiotherapy session after surgery until their discharge from hospital, which is expected to comprise one 10 minute session per day for 3-5 days.
  During each session, child participants will rate their anxiety, perceived pain and feedback any feelings about the experience.
  Interventions: Device: Immersive Virtual Reality Lower Limb and Knee Rehabilitation
- Occupational Therapist perceptions of the effectiveness of the IVR (Other): She recruited the patients, gave out devices, administered the outcome measures and provided us with feedback about their experience with the VR game.
  At the end of the trial, an interview (10 minutes) with the OT was conducted by a research nurse.
  Interventions: Device: Immersive Virtual Reality Lower Limb and Knee Rehabilitation

INTERVENTIONS:
Device: Immersive Virtual Reality Lower Limb and Knee Rehabilitation — Patients wore a VR headset while undergoing their rehabilitation session

SUMMARY:
Patients who have undergone lower limb or knee surgery are often required to participate in rehabilitative exercises to regain or maximise movement and function in the affected leg. Physiotherapy interventions for rehabilitation can be painful, uncomfortable, and tedious, reducing compliance and limiting the movement and function achieved by the patient.

Clinical studies have reported improvements in pain, compliance and outcomes by incorporating Virtual Reality (VR) into care. Evidence suggests that more Immersive VR (IVR) is effective in rehabilitation, while being cost-effective, with few adverse side-effects. Previous research by this team with adult burn patients and paediatric upper limb rehabilitation patients indicate that IVR could help reduce pain, increase compliance and improve care experiences and outcomes.

The objective of the study is to investigate the feasibility and perceived impact of the Immersive Virtual Reality (IVR) intervention as a tool in physiotherapy rehabilitation for children (aged 11-16) after lower limb or knee surgery.

DETAILED DESCRIPTION:
The study will take the form of feasibility and proof of concept trial using IVR as a physiotherapy rehabilitation tool following lower limb or knee surgery for children (aged 11 - 16). It will examine the feasibility, acceptability, usability, and efficacy of the IVR system from the perspectives of the children, parents and staff. The mixed-method approach (collecting quantitative and qualitative data):

Assess changes in anxiety, pain and movement during daily physiotherapy rehabilitation sessions after surgery and before discharge from hospital, based on:

* Child's anxiety ratings before physiotherapy
* Child's pain ratings after physiotherapy
* Practitioner's ratings of movement during physiotherapy Assess child, parent / carer and staff perceptions of and satisfaction with IVR as a tool to enhance the experience and outcomes of physiotherapy.

Assess the perceptions of therapeutic and clinical staff on the viability of the IVR as a tool for assisting in rehabilitation physiotherapy in the hospital setting.

Procedure Before consent is taken, child participants will be offered a 5 minute exposure to the HMD IVR equipment and another similar game, to familiarise themselves with the equipment, check there are no problems, and avoid unnecessary distractions and confusion during the IVR scenario itself. Patients will then use the IVR during each physiotherapy session after surgery until their discharge from hospital, which is expected to comprise one 10 minute session per day for 3-5 days. During each session, child participants will rate their anxiety, perceived pain and feedback any feelings about the experience. Physiotherapists will record the range of movement and strength using standardised measures to check for improvements.

Qualitative feedback will be gathered through interviews with children, their parents, and practitioners, focusing on experiences, satisfaction, effectiveness, acceptability, and practicality of the IVR intervention. Further feedback on IVR usability will be obtained from practitioners.

Data Analyses Descriptive statistics for anxiety, pain and movement collected before, during and after physiotherapy sessions will be calculated. Repeated measures analyses will be conducted to assess changes over time in each outcome.

Interpretive analyses will be conducted to establish whether demographic differences influence dependent variables.

Findings for anxiety, pain and movement under IVR and for SUS (usability scale) ratings will also be compared with pre-existing norm-related evidence and other relevant published clinical outcomes from physiotherapy studies. However, in this small sample, statistical analyses will be treated tentatively. Future larger scale work will strengthen any tentative findings made from this small-scale feasibility study.

Qualitative data from all interviews will be collated and analysed for themes which address the aims of the study using established thematic analysis processes. This will involve a process of careful reading, coding and comparison in order to identify important patterns in the data, focused on answering the aims of the study. Themes will be generated based upon the analysis process, which will be discussed and refined within the research team. Data will be stored, organised and analysed in NVivo.

ELIGIBILITY:
Inclusion Criteria:

* aged 11-16.
* able to speak and understand English.
* receiving physiotherapy rehabilitation treatment as an inpatient following lower limb or knee surgery, in order to restore or improve movement and function.

Exclusion Criteria:

* - Injuries to the face or head that could hinder the correct positioning of the headset or pose an infection risk
* A learning impairment that could hinder the understanding of the task
* A history of severe motion sickness or vertigo.
* Mental health problems

In order to avoid unnecessary psychological or physical distress, it is expected that we will exclude those with acute mental health symptoms as assessed by clinicians, where the use of VR might be contraindicated.

Children with mild, well controlled mental health problems will not be excluded from the study, as long as parents, child, and clinicians are in agreement. VR can occasionally cause dizziness or nausea in individuals with motion sickness, and although designed to be as enjoyable as possible, activities in the VR may cause anxiety in those with vertigo. These issues will be identified in the information sheets and discussed with parents.

Ages: 11 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 15 (Actual)
Dates: Start 2021-12-12 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
Ratings of child participant's pre physiotherapy anxiety | 3-5 days
  Child participant complete the Generalised Anxiety Disorder Assessment (GAD-7) scale measure in the data collection booklet in clinic The GAD-7 originates from Spitzer RL, Kroenke K, Williams JB, et al; A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. GAD-7 © Pfizer Inc. all rights reserved; used with permission.
  The GAD-7 score is calculated by assigning scores of 0, 1, 2, and 3, to the response categories of 'not at all', 'several days', 'more than half the days', and 'nearly every day', respectively, and adding together the scores for the seven questions.Scores of 5, 10, and 15 are taken as the cut-off points for mild, moderate and severe anxiety, respectively.
Ratings of child participant's movement during physiotherapy sessions: Goniometer (Standard BASELINE® 12-inch) | 3-5 days
  Goniometer device (Standard BASELINE® 12-inch plastic goniometer, (Model 12-1000-Fabrication Enter- prises, Inc: White Plains, New York) was used by the clinical staff before and after the patient's rehabilitation to document the initial and subsequent range of motion, evaluate their progress and to determine the level of disability. We used the goniometer, to assess the physical therapy effectiveness of the VR rehabilitation and to personalize the system's range of motion for each patient. We examined the differences between a range of movements limb join (flexion, extension, abduction, and adduction) before and after the VR rehabilitation. The greater the range of movement the better.
Ratings pain of child participant's post physiotherapy | 3-5 days
  Child participant will complete the The visual analog scale (VAS) scale measure in the data collection booklet in clinic. The VAS is a validated, subjective measure for acute and chronic pain. Scores rom 0-100 are based on self-reported measures of symptoms that are recorded with a single handwritten mark placed at one point along the length of a 10-cm line that represents a continuum between the two ends of the scale-"no pain" on the left end (0 cm) of the scale and the "worst pain" on the right end of the scale (10 cm).
  *Delgado, D. A., Lambert, B. S., Boutris, N., McCulloch, P. C., Robbins, A. B., Moreno, M. R., & Harris, J. D. (2018). Validation of digital visual analog scale pain scor
Interviews with child and parent participant | 3-5 days
  Semi-structured interviews were conducted by the research by zoom with patients and parents after the IVR rehabilitation at-home trial. Four closed ten-point Likert questions provided a quantitative measure of the perceived ease or difficulty of use, pain levels and enjoyability of the IVR system. Open-ended questions provided qualitative data relating to difficulty, pain and enjoyability, and participant attitudes towards the IVR system and its future deployment. Another semi-structured interview was conducted with the OT by the research nurse in person at the end of the trial to explore her attitudes towards the IVR system and future VR deployment. Both interviews were recorded, transcribed and anonymised.
System Usability Scale (SUS) results | 3-5 days
  System Usability Scale SUS) is a quantitative scale to measure system usability was completed by patients after the IVR rehabilitation at-home trial. It consists of a 10 item with 5-point response options from Strongly agree to Strongly disagree (Brooke, 1996). The scale evaluates the perceived ease of use (a single dimension). However, recent research shows that items 4 and 10 could provide the learnability dimension. Score contribution of each item was coded from 0 to 4 (items with positive words 1, 3, 5, 7 and 9; items with negative words 2, 4, 6, 8 and 10), and the sum of the contributions of the item scores was multiplied by 2.5 to obtain the overall SUS score (0 to 100). Scores were analysed above or below the standard mean score of 68. A score close to 100 was considered good usability of the system.

CONTACTS AND LOCATIONS:
Overall Officials: Ivan Phelan, Principal Investigator — Sheffield Hallam University
Locations (1):
- Ivan Phelan, Sheffield, South Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No